CLINICAL TRIAL: NCT01769625
Title: Prostaglandin Inhibition to Prevent Breast Cancer
Brief Title: Changes in Biomarkers Using Prostaglandin Inhibitors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Principal Investigator, Edward Sauter, MD, PhD, M.H.A, The University of Texas Health Science Center at Tyler
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 200807-001
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Biomarker Change Linked to Breast Cancer
Keywords: breast; high risk women; biomarkers; vitamin D
MeSH Terms: interventions — Celecoxib; Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- placebo & cholecalciferol 400 IU (Placebo Comparator): In this arm, the placebo is in place of celecoxib and the current RDA for cholecalciferol is used the control of the cholecalciferol higher dose.
  Interventions: Drug: placebo/celecoxib 400 mg and cholecalciferol 400 IU/cholecalciferol 2,000 IU
- placebo & cholecalciferol 2,000 IU (Active Comparator): Placebo & cholecalciferol 2,000 IU
  Interventions: Drug: placebo/celecoxib 400 mg and cholecalciferol 400 IU/cholecalciferol 2,000 IU
- celecoxib 400mg & cholecalciferol 2,000 IU (Experimental): celecoxib 400 mg & cholecalciferol2,000 IU
  Interventions: Drug: placebo/celecoxib 400 mg and cholecalciferol 400 IU/cholecalciferol 2,000 IU

INTERVENTIONS:
Drug: placebo/celecoxib 400 mg and cholecalciferol 400 IU/cholecalciferol 2,000 IU — Take 1 capsule from each bottle (1 bottle containing either placebo/celecoxib and 1 bottle containing either cholecaliferol 400 IU/cholecaliferol 2,000 IU) for 30 days
  Other Names: celecoxib (Celebrex); cholecalciferol (vitamin D); placebo (empty capule inside empty capsule

SUMMARY:
This is a biomarker study with the goal of measuring changes in proteins and gene methylation. This study is not intended for use in diagnosing, mitigating, treating, curing, or preventing disease.

The purpose of this study is to determine if Vitamin D (cholecalciferol) alone and in combination with celecoxib (Celebrex, a non-steroidal anti-inflammatory drug, or NSAID), act together to decrease breast cancer risk by their effect on certain biological indicators (biomarkers) of breast cancer risk (called PGE2, COX-2, and 15-PGDH) and cell changes in the breast.

DETAILED DESCRIPTION:
This is a biomarker study with the goal of measuring changes in protein and rna expression. This study is not intended for use in diagnosing, mitigating, treating, curing, or preventing disease.

66 women at normal risk for developing breast cancer will be recruited and enrolled. 22 women will be randomized into each arm, with anticipation of 2 women in each group will not be evaluable, leaving 20 in each group for evaluation.

A combination of vitamin D and celecoxib act synergistically to decrease breast cancer risk by decreasing cell proliferation in the mammary epithelium through their action on prostaglandin synthesis and metabolism.

Specific Aims:

-Evaluate vitamin D metabolism, through the measurement of CYP24 in the breast.

2-Evaluate breast specific levels of vitamin D and celecoxib, and assess if the levels of these compounds correlate with response to markers which influence prostaglandin synthesis and metabolism. Additionally, in women without active breast cancer , we will determine the effect of vitamin D, with or without celecoxib, on 1) PG synthesis and metabolism, through the measurement of PGE2, COX-2 and 15-PGDH in the breast, 2) proliferative activity in the breast,, and 3) circulating levels of vitamin D and celecoxib, to determine if levels of these compounds correlate with response to markers of PG production, metabolism, or cell proliferation.

ELIGIBILITY:
Inclusion Criteria:

* Woman >18 years old
* Healthy women who are at normal risk for developing breast cancer
* ECOG Performance Status score 0-1
* Premenopausal women must not be pregnant

Exclusion Criteria:

* History of bilateral mastectomy, or bilateral breast irradiation
* Significant medical or psychiatric problems making the participant a poor candiate
* Evidence of excess use of narcotics or drug dependency
* Have been pregnant and lactating in the past 2 years
* Significant history of peptic ulcer disease or upper gastrointestinal bleeding
* History of severe congestive heart failure that requires hospitalization or intervention
* History of asthma requiring medication for treatment
* Allergy to sulfonamides or NSAID medications
* History of myocardial infarction or stroke
* Currently on Coumadin
* Currently on Tamoxifen (nolvadex),Evista (raloxifene), Femara (letrozole), Arimidex (anastrozole), or Aromasin (exemestane)
* Undergone prior subaeolar breast surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-01; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
PG synthesis and metabolism, through the measurement of PGE2, COX-2 and 15-PGDH in the breast | approximately 30 days
  This will be measured from both baseline and completion samples
  1. PG synthesis and metabolism, through the measurement of 15-PGDH, COX-2, and PGE2 in the breast
  Rationale: 1,25(OH)2D, the active form of vitamin D, has been shown in vitro to decrease PGE2 both by interfering with its production and by increasing its breakdown, leading to lower cell proliferation. Celecoxib potentiated the antiproliferative effect, allowing a much lower dose of each agent when used in combination than in isolation.

SECONDARY OUTCOMES:
proliferative activity in the breast and circulating levels of vitamin D and celecoxib, to determine if levels of these compounds correlate with response to markers of PG production, metabolism, or cell proliferation. | approximately 30 days
  This will be measured from both baseline and completion samples.
  2. Proliferative activity in the breast, as measured by MD cell morphology
  Rationale: Both MD and NAF contain ductal epithelial cells, but MD samples contain more cells for cytologic review than NAF. Findings on MD cytology correlate with likelihood of breast cancer, NAF cytology relates to breast cancer risk and improves risk stratification, and bioactive food components can alter NAF cytology

CONTACTS AND LOCATIONS:
Overall Officials: Edward R. Sauter, MD, PhD, M.H.A, Principal Investigator — University of North Dakota
Locations (1):
- University of North Dakota, Grand Forks, North Dakota, United States